CLINICAL TRIAL: NCT02501291
Title: Thalidomide in Inducing and Maintaining Remission of Crohn's Disease
Brief Title: Thalidomide in Treating Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ren Mao, MD,PhD, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBD201501
Record Dates: First submitted 2015-05-20; First posted 2015-07-17 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide (Experimental): Thalidomide was administered at a daily dose of 50 mg to the patients. Dosage adjustment of thalidomide from 25mg daily to 100mg daily was tailored individually according to patients' tolerance to thalidomide. To minimize the sedative effect of thalidomide, the investigators recommended patients take a single dose of the study drug in the evening before bedtime.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
Crohn's disease (CD) is a chronic gastrointestinal inflammatory disease characterized by relapse and progression. The incidence and prevalence of IBD are increasing in different regions around the world, indicating its emergence as a global disease. Though modern medical therapies including immunomodulators and biologic agents have revolutionized treatment of CD, the occurrence of steroids-dependence and resistance or intolerance to medical therapy is quite common. The limitation of present therapeutic management and the high expense of biologic agents leads to the treatment of CD become "refractoriness". The occurrence rate of steroids-dependence and resistance or intolerance to thiopurine therapy is quite high during the course of CD. Approximately 38% of cases required surgery within 10 years. Therefore, the management of such refractory CD remains a great therapeutic challenge for clinicians.

Thalidomide is an oral agent that has immunomodulatory, antiangiogenic and TNF(tumor necrosis factor)-a- suppressing effects. The potential role for thalidomide in the treatment of refractory paediatric and adult CD has been investigated in more and more small open-label studies and retrospective case series. Recently, a randomized controlled trial showed thalidomide improved clinical remission at 8 weeks of treatment and longer-term maintenance of remission in pediatric refractory CD. Gerich et al reported in a retrospective study that thalidomide improved long-term outcomes among 37 refractory CD adults followed up for a median of 58 months. However, the dose of thalidomide used in these studies ranged from 50mg/d to 150mg/d, and the occurrence rate of side effects reported variously but all quite high. The side effects related to the dose of thalidomide were the major concerns of using it in CD. Moreover, the effect of thalidomide on endoscopic response including mucosal healing which is a more objective and important outcome in CD was rarely reported. Therefore the aim of this study is to investigate the efficacy on clinical and endoscopic response and the adverse effects of using low-dose thalidomide in active adult CD patients.

ELIGIBILITY:
Inclusion Criteria:

A CDAI score greater than 150 at baseline was required for inclusion .(1) steroid-dependent: unable to reduce steroids below the equivalent of prednisone 10 mg/day (or budesonide below 3 mg/day) within 3 months of starting steroids, or who have a relapse within 3 months of stopping steroids.(2) thiopurines-non-responsive: active disease or clinical relapse despite administration of azathioprine (1.5-2 mg per kg per day) or 6-mercaptopurine (0.75-1.5 mg per kg per day) for 4 months. (3) thiopurines- intolerant: intolerance to or adverse events of thiopurines.

The exclusion criteria were (1) isolated L4 CD; (2) disease including symptomatic stenosis of intestine or abdominal abscess requiring immediate surgery; (3) Current or past history of malignancy or organ transplantation; (4) Serious infections within 3 months; (5) Previous history of neuropathy or symptoms of neuropathy or abnormal electromyography prior to thalidomide; (6) infliximab treatment in the previous 8 weeks; (7) progressive or uncontrolled renal, hepatic, hematological, pulmonary and cardiac disease and（8）ongoing pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Clinical remission | 8 weeks
  Clinical remission is defined as CDAI (Crohn's disease activity index) less than 150.

SECONDARY OUTCOMES:
clinical response and endoscopic efficacy | 24 weeks
  Clinical response was defined as a decrease in CDAI score of ≥100 points from baseline. Endoscopic efficacy was reassessed by ileocolonoscopy at week 24. Endoscopic outcome measures included endoscopic response (decrease in CDEIS score >5 points from baseline of CDEIS of 6 or more), complete remission (CDEIS score <3) and mucosal healing (no ulcer)response was defined as a decrease in CDAI score of ≥100 points from baseline. Endoscopic efficacy was reassessed by ileocolonoscopy at week 24. Endoscopic outcome measures included endoscopic response (decrease in CDEIS score >5 points from baseline of CDEIS of 6 or more), complete remission (CDEIS score <3) and mucosal healing (no ulcer)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Lazzerini M, Martelossi S, Magazzu G, Pellegrino S, Lucanto MC, Barabino A, Calvi A, Arrigo S, Lionetti P, Lorusso M, Mangiantini F, Fontana M, Zuin G, Palla G, Maggiore G, Bramuzzo M, Pellegrin MC, Maschio M, Villanacci V, Manenti S, Decorti G, De Iudicibus S, Paparazzo R, Montico M, Ventura A. Effect of thalidomide on clinical remission in children and adolescents with refractory Crohn disease: a randomized clinical trial. JAMA. 2013 Nov 27;310(20):2164-73. doi: 10.1001/jama.2013.280777. PMID 24281461
- [Result] Gerich ME, Yoon JL, Targan SR, Ippoliti AF, Vasiliauskas EA. Long-term outcomes of thalidomide in refractory Crohn's disease. Aliment Pharmacol Ther. 2015 Mar;41(5):429-37. doi: 10.1111/apt.13057. Epub 2014 Dec 15. PMID 25511905